CLINICAL TRIAL: NCT02679053
Title: Aerobic Exercise as add-on Treatment for Inpatients With Depression: Effects and Biomarkers
Brief Title: Aerobic Exercise as add-on Treatment for Inpatients With Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Collaborators: Psychiatric Hospital of the University of Basel (Other); University of Basel (Other); Solothurner Spitäler AG (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: EKBB 62/13
Record Dates: First submitted 2016-01-26; First posted 2016-02-10 (Estimated); Last update posted 2017-04-11 (Actual); Status verified 2017-04

CONDITIONS: Depression
MeSH Terms: conditions — Depression | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Exercise (IG) (Experimental): Aerobic exercise three times per week on indoor bicycles at 60 to 75% of maximal heartrate aiming at a weekly total of 17.5kcal/kg bodyweight for 6 consecutive weeks. The exercise will take place under supervision. At the end of every week physical fitness is evaluated by the queens step test.No other activities with moderate or high intensity are allowed throughout the intervention time.
  Interventions: Behavioral: Aerobic exercise
- Control (CG) (Placebo Comparator): Basic stretching and mobilisation program 3 times per week each for approx. 40 minutes, also under supervision for 6 consecutive weeks. At the end of every week physical fitness is evaluated by the queens step test.At the end of every week physical fitness is evaluated by the queens step test.No other activities with moderate or high intensity are allowed throughout the intervention time.
  Interventions: Behavioral: Placebo control

INTERVENTIONS:
Behavioral: Aerobic exercise
  Arms: Exercise (IG)
Behavioral: Placebo control
  Arms: Control (CG)

SUMMARY:
The aim of the study is to evaluate the effect of 6 weeks of aerobic endurance exercise as adon treatment for moderately to severely depressed inpatients. Endpoints are symptom severity, psychological variables, cognitive symptoms, sleep, hypothalamic-pituitary-adrenal axis (HPA-axis), Brain-derived neurotrophic factor (BDNF) and heartrate variability (HRV).

Amendment 1 (Nov. 2016): additional evaluation of TNF-alpha at baseline, +2 weeks and post (+6weeks) in already existing blood samples.

DETAILED DESCRIPTION:
Patients are randomly assigned to the intervention group (IG) or control group (CG). The IG will train three times per week on indoor bicycles at 60 to 75% of maximal heartrate aiming at a weekly total of 17.5kcal/kg bodyweight for 6 consecutive weeks. The exercise will take place under supervision. CG will absolve a basic stretching and mobilisation program 3 times per week, also under supervision for 6 consecutive weeks. At the end of every week physical fitness is evaluated by the queens step test. No other activities with moderate or high intensity are allowed throughout the intervention time.

All patients will participate in the multimodal treatment program of the depression ward, which includes pharmacotherapy, psychotherapy and specialized therapies such as art therapy and ergotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Inpatient treatment on the Depression ward
* International Classification of Diseases (ICD)-10: F32, F33 or F31
* HDRS-17>16 Points
* written informed consent

Exclusion Criteria:

* Any physical condition that prohibits endurance exercise
* 3 or more cardiovascular risk factors (hypertonia, family history, smoking, hypertriglyceridemia, diabetes)
* pathological ECG
* BMI > 35 kg/m2
* Pregnancy
* acute suicidal Ideation
* comorbid substance dependence (except nicotine)
* Major comorbid psychiatric disorder
* regular high intensity exercise prior to treatment

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 49 (Actual)
Dates: Start 2013-10; Primary Completion 2016-02 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Depressive Symptoms self rated | Baseline (pre), 1 week, 2 weeks, 6 weeks (post), 6 months (followup)
  Change in Score of Hamilton Depression Rating Scale (HDRS-17) from baseline until 6 months follow-up
Depressive Symptoms physician rated | Baseline (pre), 1 week, 2 weeks, 6 weeks (post), 6 months (follow-up)
  Change in Score of Beck Depression Inventory (BDI) from baseline until 6 months follow-up

SECONDARY OUTCOMES:
Cortisol awakening response (CAR) | Baseline (pre), 2 weeks, 6 weeks (post), 6 months (follow-up)
  Change of Salivary cortisol increase (Area under the curve, measured at awakening, +10, +20 and +30 minutes) from baseline until 6 months follow-up
Brain derived neurotrophic factor (Serum-BDNF) | Baseline (pre), 2 weeks, 6 weeks (post), 6 months (followup)
  Change of Serum-BDNF
Sleep (Subjective sleep Quality) | Baseline (pre), 6 weeks (post), 6 months (followup)
  Change of Score of Pittsburgh sleep quality index (PSQI) from baseline until follow-up
Sleep (Polysomnography) | Baseline (pre), 6 weeks (post)
  Change in sleep stages between baseline and follow-up
Cognition | Baseline (pre), 6 weeks (post), 6 months (followup)
  Change in performance in Executive functions (alertness, working memory, flexibility, go/nogo, divided attention) measured by "Testbatterie zur Aufmerksamkeitsprüfung" (TAP)
Social stress - cortisol | Baseline (pre), 6 weeks (post)
  Change of Salivary cortisol-course (Area under the curve) during Trier Social Stress Test (TSST)
Social stress - heartrate | Baseline (pre), 6 weeks (post)
  Change of heartrate-course during Trier Social Stress Test (TSST)
Psychological symptoms | Baseline (pre), 6 weeks (post), 6 months (follow-up)
  Change of scores in Symptom Checklist (SCL-90R) from baseline until follow-up
Mental Toughness | Baseline (pre), 6 weeks (post), 6 months (followup)
  Change in score in Mental Toughness Questionnaire (MTQ18)from baseline until follow-up
Physical activity | Baseline (pre), 6 months (follow-up)
  Change of weekly physical activity as self reported by the International Physical Activity Questionnaire - Short Version (IPAQ-short)
Sleep related personality traits | Baseline (pre), 6 weeks (post), 6 months (followup)
  Change in Focussing and Rumination subscores of the "Fragebogen zur Erfassung von Persönlichkeitsmerkmalen Schlafgestörter" (FEPS II)
Body Mass Index (BMI) | Baseline (pre), 6 weeks (post), 6 months (followup)
  Change(BMI)
Resting Heartrate (HR) | Baseline (pre), 6 weeks (post), 6 months (followup)
  Change of HR
Blood Pressure (BP) | Baseline (pre), 6 weeks (post), 6 months (followup)
  Change of BP
TNF-Alpha (additional value assessed/Amendment 1) | Baseline (pre), 2 weeks (post), 6 weeks (post)
  Change of TNF-alpha

CONTACTS AND LOCATIONS:
Overall Officials: Christian Imboden, MD, Dr., Principal Investigator — Solothurner Spitäler AG
Locations (2):
- Switzerland (2):
  - Psychiatric University Hospital, Basel, Basel
  - Psychiatric Services Solothurn, Solothurn, Canton of Solothurn

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Imboden C, Gerber M, Beck J, Eckert A, Puhse U, Holsboer-Trachsler E, Hatzinger M. Effects of Aerobic Exercise as Add-On Treatment for Inpatients With Moderate to Severe Depression on Depression Severity, Sleep, Cognition, Psychological Well-Being, and Biomarkers: Study Protocol, Description of Study Population, and Manipulation Check. Front Psychiatry. 2019 Apr 25;10:262. doi: 10.3389/fpsyt.2019.00262. eCollection 2019. PMID 31073292